CLINICAL TRIAL: NCT04207164
Title: Translation, Cross-culture Adaption of Foot Functional Index Revised, Short Version (FFI-RS) Into Norwegian. Testing of Psychometric Properties.
Brief Title: Translation and Psychometric Testing of the Norwegian Foot Functional Index Revised, Short Version.
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Mørk, Physical Therapist, Oslo University Hospital
Other Study IDs: 1045762
Record Dates: First submitted 2019-11-01; First posted 2019-12-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Foot Diseases; Plantar Fascitis
Keywords: Foot Functional Index revised,; Translation and cultural adaption; Reliability; Validity; Responsiveness
MeSH Terms: conditions — Foot Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to translate into Norwegian and cross-culturally adapt the Foot Functional Index- revised, short form (FFI-RS) according to international guidelines. Furthermore, the reliability and the validity, responsiveness as well as floor and ceiling effect of the Norwegian version of the FFI-RS will be determined.

DETAILED DESCRIPTION:
Foot Functional Index, revised short form is a foot specific patient reported outcome measurement (PROM) which covers pain, stiffness, activity limitations, disability as well as psychosocial issues.

The aim of this study is to translate into Norwegian and cross-culturally adapt Foot Functional Index revised, short form (NFFI-RS). Furthermore, the reliability, validity, interpretability and responsiveness will be determined.

The Department of Physical Medicine and Rehabilitation at Oslo University Hospital has an ongoing double blind, randomized sham-controlled trial (RCT) comparing the effect of radial extracorporeal shock wave therapy (rESWT), sham rESWT, standardized exercise program and usual care for patients with longstanding plantar fasciopathy (NCT03472989). The testing of the psychometric properties of the NFFI-RS will include totally hundred patients, both from the mentioned RCT as well as patients with other foot diagnosis recruited from our department.

The translation of the original FFI-RS into Norwegian has been done following the official guidelines.

In the test-retest study fifty patients will complete the NFFI-RS at a one week interval.

Smallest detectable change, measurement error, floor and ceiling effects as well as internal consistency will be calculated by using the baseline data. To decide the construct validity we will test the various hypothesis at baseline.

To calculate the responsiveness and the minimal clinically important change three months data will be assessed. Patient Global Impression of Change Scale will be used to assess the minimal clinically important change and responsiveness of the NFFI-RS with ROC and AUC analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain localized in the foot
* Patients understanding oral and written Norwegian

Exclusion Criteria:

* Patients without pain in the foot
* Patients not understanding oral and written Norwegian

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with foot pain attending the Department of Physical Medicine and Rehabilitation at Oslo University Hospital (OUS), Norway will be included. Some of the patients will have the diagnosis Plantar Fasciopathy (PF) and is a part of the ongoing RCT from the same department at OUS: "The effectiveness of radial extracorporeal shock wave therapy (rESWT), sham rESWT, standardised exercised exercise programme or usual care for patients with plantar fasciopathy." (NCT03472989)(2017/1325 Regional Comimittee for Medical and Health Research Ethics,Norway).
  Rest of the study population will be patients with othe foot complaints.
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Foot Functional Index revised short version ( FFI-RS) | Baseline, 1 week, 3 months
  FFI-RS is a foot specific pain and function score. We will evaluate the reliability of the FFI-RS by testing the internal consistency (Cronbach's Alpha). Furthermore test-retest will be done with a second FFI-RS recording after one week (weighted Kappa). We will evaluate construct validity with other instruments (RAND-12 and NRS). To test the responsiveness of FFI-RS, we will evaluate the change in FFI-RS from baseline to 3 months with Patient Global Impression of Change score.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | Baseline
  Change in heel pain (during Activity last week). NRS is a patient reported pain intensity scale ranging from 0 (no pain) to 10 (worst possible pain). NRS will by used for evaluating the construct validity of FFI-RS.
RAND-12 | Baseline
  Health related quality of life (12 items). RAND-12 will be used for evaluating the construct validity of FFI-RS.
Patient Global Impression Of Change Scale (PGIC) | 3 months
  7-point scale ranging from "very much improved" to "very much worse". PGIC will be used for evaluating the responsiveness of FFI-RS.

CONTACTS AND LOCATIONS:
Overall Officials: Aasne F Hoksrud, MD, PhD, Study Director — Oslo University Hospital, Department of Physical Medicine and Rehabilitation
Locations (1):
- Oslo University Hospital, Department of Physical Medicine and Rehabilitation, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Budiman-Mak E, Conrad KJ, Roach KE. The Foot Function Index: a measure of foot pain and disability. J Clin Epidemiol. 1991;44(6):561-70. doi: 10.1016/0895-4356(91)90220-4. PMID 2037861
- [Result] Budiman-Mak E, Conrad K, Stuck R, Matters M. Theoretical model and Rasch analysis to develop a revised Foot Function Index. Foot Ankle Int. 2006 Jul;27(7):519-27. doi: 10.1177/107110070602700707. PMID 16842719
- [Result] Hays RD, Morales LS. The RAND-36 measure of health-related quality of life. Ann Med. 2001 Jul;33(5):350-7. doi: 10.3109/07853890109002089. PMID 11491194
- [Result] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Result] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Result] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Derived] Mork M, Hoksrud AF, Soberg HL, Zucknick M, Heide M, Groven KS, Roe C. "Psychometric properties of the Norwegian foot function index revised short form". BMC Musculoskelet Disord. 2022 May 3;23(1):416. doi: 10.1186/s12891-022-05374-x. PMID 35505330